CLINICAL TRIAL: NCT01486953
Title: Phase 4 Study of Desflurane and Sevoflurane That Affect Pulmonary Mechanics During Minimally Invasive Repair of Pectus Excavatum
Brief Title: Pulmonary Mechanics During Minimally Invasive Repair of Pectus Excavatum
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jeong Eun Kim, Clinical Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: pectus-study
Record Dates: First submitted 2011-11-26; First posted 2011-12-07 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Pectus Excavatum
Keywords: respiratory resistance; lung compliance; desflurane; sevoflurane
MeSH Terms: conditions — Funnel Chest | interventions — Desflurane; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sevoflurane (Active Comparator): Anesthesia with sevoflurane
  Interventions: Drug: Sevoflurane
- Desflurane (Experimental): Anesthesia with desflurane
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Desflurane — Using random numbers, patients were divided into two groups to receive either sevoflurane or desflurane. After induction of anesthesia and intubation, the patient's lungs were ventilated in constant-flow VCV mode by an anesthetic Ventilator (Datex-Ohmeda, GE healthcare, Finland). Ventilator settings were tidal volume 10 ml/kg, inspiratory:expiratory (I:E) ratio 1:1.5, inspired oxygen concentration (FiO2) 0.5 with air, and 3 L/min of inspiratory fresh gas flow. End-inspiratory pause was set 20% of total breathing cycle. Positive end-expiratory pressure (PEEP) was not used. Respiratory rate was adjusted to maintain an end-tidal CO2 pressure of 33-35 mmHg. Patients received desflurane 6-7% for maintenance of anesthesia.
  Arms: Desflurane
Drug: Sevoflurane — Using random numbers, patients were divided into two groups to receive either sevoflurane or desflurane. After induction of anesthesia and intubation, the patient's lungs were ventilated in constant-flow VCV mode by an anesthetic Ventilator (Datex-Ohmeda, GE healthcare, Finland). Ventilator settings were tidal volume 10 ml/kg, inspiratory:expiratory (I:E) ratio 1:1.5, inspired oxygen concentration (FiO2) 0.5 with air, and 3 L/min of inspiratory fresh gas flow. End-inspiratory pause was set 20% of total breathing cycle. Positive end-expiratory pressure (PEEP) was not used. Respiratory rate was adjusted to maintain an end-tidal CO2 pressure of 33-35 mmHg. Patients received sevoflurane 2-2.5% for maintenance of anesthesia.
  Arms: sevoflurane

SUMMARY:
The aim of the current study was to compare the effects of sevoflurane and desflurane on respiratory mechanics in patients undergoing repair of pectus excavatum.

DETAILED DESCRIPTION:
The minimally invasive technique for pectus excavatum repair was introduced by Nuss and colleagues using a metal bar to lift the depressed chest wall. This surgical procedure is usually done under general anesthesia with tracheal intubation. After inserting metal bar into the chest wall, decreased lung compliance was shown. Previous studies demonstrated that administering desflurane during anesthesia resulted in marked increases in respiratory mechanical parameters, especially in the children with airway susceptibility. Our primary hypothesis was that desflurane would cause an increase in respiratory resistance and a decrease in lung compliance compared to sevoflurane during repair of pectus excavatum.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Pectus Excavatum
* undergoing minimally invasive repair

Exclusion Criteria:

* younger than 15 year old
* history of upper respiratory tract infection within recent 2 weeks
* asthma
* chronic obstructive pulmonary disease
* previous treatment with bronchoactive drugs (B-agonist or antagonist, theophyline, anticholinergics and corticosteroid)
* history of neurological deficits

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
pulmonary mechanics | within the 2 hours during the surgery
  respiratory resistance dynamic and static lung compliance

SECONDARY OUTCOMES:
complication | within 72 hours after sugery
  bronchospasm dyspnea pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Eun Kim, M.D, Ph.D, Principal Investigator — Department of Anesthesiology, The Catholic University of Korea, Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea